CLINICAL TRIAL: NCT07104552
Title: Comparing Short to Standard Amoxicillin Course for Erysipelas: a Non-inferiority Randomized Controlled Trial
Brief Title: Comparing Short to Standard Amoxicillin Course for Erysipelas
Acronym: SHAREII
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P150924; 2024-515306-61-00 (EU CTIS Number)
Record Dates: First submitted 2025-07-29; First posted 2025-08-05 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-07

CONDITIONS: Erysipelas
Keywords: dermatology; Erysipela; amoxixillin; general practitioner
MeSH Terms: conditions — Erysipelas

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amox5Days (Experimental): Amoxicillin 50 mg/kg for five days
  Interventions: Drug: Course of amoxicillin
- Amox10Days (Active Comparator): Amoxicillin 50 mg/kg for ten days
  Interventions: Drug: Course of amoxicillin

INTERVENTIONS:
Drug: Course of amoxicillin — Oral amoxicillin per os at 50 mg/kg/day

SUMMARY:
Erysipelas is an acute streptococcal skin infection, primarily affecting the lower limbs and easily diagnosed. In 2000, the French expert consensus conference validated oral amoxicillin at 3 to 4.5 gr per day for 10 to 20 days as a standard treatment, despite the lack of full market approval for erysipelas treatment. In practice, general practitioners (GPs) typically prescribe amoxicillin for around 10 days. In 2019, the Haute Autorité de Santé (HAS), one of the national French Health Authorities, recommended a 7-day antibiotic course for erysipelas, while no RCT was available. Reducing the length of antibiotic courses during acute infections is challenging but necessary to lower therapeutic costs, reduce the risk of bacterial resistance, and improve patient adherence to treatment.

This RCT aims to validate the use of a short course, specifically 5 days, of oral amoxicillin at 50 mg/kg to treat erysipelas, demonstrating its non-inferiority compared to the standard course. The primary objective is to show that a short course (5 days) of amoxicillin at 50 mg/kg is non-inferior to the usual course (10 days) in achieving complete erysipelas remission by day 12 ± 2. The primary end point will be confirmed by a central independent committee, blinded to the intervention received, using photos and clinical data.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years
* Affiliated to a social security scheme
* Who have given written consent according to local regulatory requirements after the nature of the study has been explained to them, and prior to any protocol specific procedures being performed,
* Clinical signs of lower limbs erysipelas ≤ 5 days defined as:

  o Warmth, erythema, edema (induration of the skin and/or subcutaneous tissue) and/or pain (NRS≤8)
* Shiver, feverish sensation or fever experienced by the patient ≤ 5 days or fever measured by the physician ≥ 38°C
* Severity score ≥ 3 scored on three criteria: edema, erythema, pain with the following scales (0= none, 1=moderate, 2=severe)
* Absence of erysipela ≤ 12 months
* Absence of blisters
* Absence of solid purpura (purple tablecloth not erasing at vitro-pressure)
* Absence of cutaneous necrosis
* Absence of crepitation (crepitation = perception identical to that of cutaneous emphysema

Exclusion Criteria:

* Allergy to ß lactam, fructose intolerance
* Weight < 40 kg or > 105 kg
* Use of oral antibiotic within 5 days (excluding one or two antibiotic intake ≤ 24 hours)
* Erysipela/Cellulitis requiring hospitalization
* Bilateral erysipela
* Abscess
* Lymphedema requiring permanent contention
* Animal bite ≤ 7 days
* HIV positive
* Patient with comorbidity: known active hepatitis, chronic kidney failure or hepatocellular insufficiency
* Patient unable to temporarily stop a long-term treatment as antibiotics or corticosteroids, or NSAIDs
* Patient under immunosuppressive or oncologic treatments ≤ 6 months
* Pregnant women or breastfeeding
* Patient under guardianship or curatorship, legal protection or protection of justice
* Participation in other Clinical Trial, interventional study, investigational study or performance study Any medical, mental, psychological or psychiatric condition considered by the investigator as compromising patient completion or understanding of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 656 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2029-01-12 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
Rate of complete remission. Complete remission is a composite outcome defined as | At day 12 +/- 2
  1. the disappearance of fever (T°≥ 38°) AND of pain, warmth tenderness erythema and edema at the site of erysipelas and for the cutaneous plaque a clinical severity score less than or equal to 1; and
  2. the absence of additional antibiotherapy for the initial condition, i.e., erysipelas/cellulitis.
  The clinical severity score corresponds to the addition of the 3 score value of pain, warmth tenderness erythema and edema.
the disappearance of fever (T°≥ 38°) | At day 12 +/- 2
  T<38°
the disappearance of pain | At day 12 +/- 2
  the pain is measured from the numerical assessment (EN). The score is graded according to the following EN values:
  * if EN = 0, this equates to score 0 (Absent)
  * If EN between 1 and 8, this corresponds to a score of 1 (Moderate)
  * IF IN > 8, this corresponds to a score of 2 (Severe)
warmth tenderness erythema at the site of erysipela | At day 12 +/- 2
  It is graded according to the following values:
  * if absent, this equates to score 0
  * If moderate, this corresponds to a score of 1
  * if severe, this corresponds to a score of 2
edema at the site of erysipela | At day 12 +/- 2
  It is graded according to the following values:
  * if absent, this equates to score 0
  * If moderate, this corresponds to a score of 1
  * If severe, this corresponds to a score of 2
Number of patients who did not receive any additional antibiotics for erysipelas/cellulitis | At day 12 +/- 2
  absence of additional antibiotherapy for erysipelas/cellulitis

SECONDARY OUTCOMES:
Rate of clinical remission: the disappearance of fever (T°≥38°) AND of pain, warmth tenderness erythema and edema at the site of erysipelas and for the cutaneous plaque a clinical severity score less than or equal to 1 at day 12+/- 2 | At day 12 +/- 2
Rate and number of patients not receiving additional antibiotherapy at day 12+/- 2 | at day 12+/- 2
Rate of recurrence is defined by the need for additional antibiotic therapy for cellulitis between day 12 and day 28+/- 2. | at day 12 and day 28+/- 2
Rate of adverse event during the treatment and the follow up periods as reported by the patient | at day 12+/- 2
Rate of clinical remission: disappearance of fever (≥38) AND pain, warmth tenderness erythema and edema at the site of erysipelas and for the cutaneous plaque a clinical severity score less than or equal to 1, without receiving additional antibiotherapy | at day 7 +/- 2

CONTACTS AND LOCATIONS:
Overall Officials: France Guyot, Study Chair — Assistance Publique Hôpitaux de Paris - DRCI